CLINICAL TRIAL: NCT07067450
Title: Adjuvant Immunotherapy Versus Observation Following Neoadjuvant Chemoimmunotherapy for Esophageal Squamous Cell Carcinoma: A Randomized Controlled Trial
Brief Title: Adjuvant Immunotherapy for Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-ESCC
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: esophageal squamous cell carcinoma; neoadjuvant chemoimmunotherapy; Adjuvant immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Immune Checkpoint Inhibitors; pembrolizumab; tislelizumab; sintilimab; camrelizumab; toripalimab; Observation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Immunotherapy Group (Experimental): For patients with non-pCR esophageal squamous cell carcinoma after neoadjuvant chemoimmunotherapy, adjuvant immunotherapy with immune checkpoint inhibitors (the same ICIs used before surgery) is administered postoperatively, once every three weeks, for a total of 15 treatments.
  Interventions: Drug: Immune Checkpoint Inhibitors ( pembrolizumab, tislelizumab, sintilimab, camrelizumab, and toripalimab)
- Observation Group (Active Comparator): For patients with non-pCR esophageal squamous cell carcinoma after neoadjuvant chemoimmunotherapy, postoperative observation is conducted without the use of any anti-tumor treatment.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors ( pembrolizumab, tislelizumab, sintilimab, camrelizumab, and toripalimab) — The immune checkpoint inhibitors used for adjuvant therapy after surgery were consistent with those used during the neoadjuvant treatment before surgery, including pembrolizumab, tislelizumab, sintilimab, camrelizumab, and toripalimab.
  Arms: Adjuvant Immunotherapy Group
Other: Observation — Postoperative observation is conducted without the use of any anti-tumor treatment.
  Arms: Observation Group

SUMMARY:
Patients with esophageal cancer still face a high risk of recurrence after receiving neoadjuvant chemoradiotherapy (nCRT) combined with radical surgery, especially for those who do not achieve pathological complete response (non-pCR). Compared with the overall non-pCR population, the subgroup with lymph node positivity has a significantly worse prognosis. The CheckMate 577 study confirmed that in patients with locally advanced resectable esophageal cancer or esophageal-gastric junction cancer, adjuvant treatment with nivolumab after nCRT significantly prolonged disease-free survival compared with placebo (median DFS: 22.4 months vs 11.0 months; HR=0.69, p<0.001).

The current research focus has expanded to the field of neoadjuvant chemoimmunotherapy, but the adjuvant treatment strategy after such therapy remains a blank slate. Given that esophageal squamous cell carcinoma (ESCC) is the predominant type of esophageal cancer in our country, it is of great clinical significance to explore adjuvant treatment strategies after neoadjuvant chemoimmunotherapy combined with radical resection.

Based on the above background, we have designed a randomized controlled trial (RCT) to evaluate the efficacy of adjuvant immunotherapy versus observation alone in patients with ESCC after neoadjuvant chemoimmunotherapy, with the hope of providing evidence-based medical evidence for this population.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Histologically confirmed esophageal squamous cell carcinoma.
* Preoperative staging of cT1b-cT2N+M0 or cT3-cT4a, any N, M0 (UICC/AJCC TNM staging, 8th edition, 2017), and treated with neoadjuvant therapy using an immunotherapy combined with a taxane and platinum regimen, followed by radical surgical resection.
* R0 resection.
* Postoperative pathological staging of ≥ypT1 and/or ≥ypN1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
* Physical examination and imaging studies completed within 4 weeks prior to randomization confirming disease-free status, with imaging studies including CT scans of the chest and abdomen.
* Normal function of major organs.
* Women of childbearing potential and men with partners of childbearing potential must agree to use effective contraception during the treatment period and for 6 months before and after the treatment period.
* Willingness of the subject to participate in the study and provision of informed consent.
* Good compliance of the subject, with the ability to follow up on efficacy and adverse events/reactions as required by the study plan.

Exclusion Criteria:

* Presence of blood-borne infectious disease human immunodeficiency virus (HIV).
* Presence of psychiatric disorders.
* History of any other malignancy within the past 5 years (except for completely cured cervical carcinoma in situ or basal cell or squamous cell carcinoma of the skin).
* Treatment in the ICU due to severe complications after radical surgery for esophageal cancer.
* Severe anastomotic stricture after surgery, requiring dilation treatment.
* Known severe allergy to any component of the study drug.
* Presence of other autoimmune diseases, or long-term systemic use of immunosuppressants or corticosteroids; the use of inhaled or topical corticosteroids or equivalent doses of adrenal corticosteroid replacement therapy is permitted.
* Active hepatitis B (HBV-DNA ≥ 2000 IU/mL or 10⁴ copies/mL), hepatitis C (positive hepatitis C antibody, and HCV-RNA above the lower limit of detection of the assay). Patients with a hepatitis B copy number ≤ 10³ copies/mL after anti-hepatitis B or C treatment may be considered for enrollment at the discretion of the principal investigator.
* Presence of any unstable systemic disease (including active uncontrolled peptic ulcer, active infection, grade 4 hypertension, unstable angina, congestive heart failure, unstable cerebrovascular disease, thromboembolic disease, hepatic, renal, metabolic diseases, or unhealed fractures, wounds as judged by the surgeon).
* Patients who are difficult to communicate with or follow up with over the long term.
* Women who are breastfeeding.
* Currently participating or planning to participate in other clinical trials.
* Other situations deemed unsuitable by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From the time of patient enrollment, up to a maximum of 2 years.
  In this study, disease-free survival (DFS) refers to the time from the start of surgery to the first occurrence of disease recurrence or metastasis. If a patient does not experience disease recurrence or metastasis during the follow-up period, their DFS is typically recorded as the time from the start of treatment to the end of follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the time of patient enrollment, up to a maximum of 5 years.
  Overall Survival (OS) refers to the time from the start of enrollment to the time of death from any cause. If a patient is still alive at the end of the study, their OS is recorded as the time from the start of the study to the end of the study.